CLINICAL TRIAL: NCT06677944
Title: Impact of Preoperative Stereotactic Partial Breast Irradiation on Treatment Response, Treatment-related Toxicity, and Cosmetic Outcomes in Early-stage Breast Cancer: A Prospective, Phase II Clinical Trial
Brief Title: Preoperative Partial Breast Irradiation in Early-Stage Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-1112
Record Dates: First submitted 2024-01-23; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Ductal Carcinoma in Situ; Invasive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative PBI (Experimental): PBI before surgery
  Interventions: Radiation: Preoperative PBI

INTERVENTIONS:
Radiation: Preoperative PBI — Preoperative PBI: 21 Gy * 1 fraction Preoperative PBI is administered within 6 weeks of the patient's initial registration, and surgery is scheduled within 8 to 12 weeks after PBI.

SUMMARY:
In the management of early breast cancer patients, postoperative radiotherapy following breast-conserving surgery has been established as the standard treatment. Over the past two decades, significant changes have occurred in radiotherapy for breast cancer, encompassing dose fractionation methods, radiotherapy techniques, and delineation of the radiation field. Hypofractionated radiotherapy has been reported in numerous randomized phase 3 studies to show equivalent tumor control rates, reduced acute side effects, and similar late side effects compared to conventional fractionation. Among hypofractionated radiotherapy approaches, particularly in early-breast cancer, accelerated partial breast irradiation (APBI) may be chosen over whole breast irradiation (WBI). This approach is based on data indicating that the majority of local recurrences in breast cancer occur around the site of the primary tumor. By targeting radiation to the involved breast region, it becomes possible to increase the dose per fraction while shortening the overall treatment duration due to the smaller radiation treatment volume. While careful patient selection is crucial, multiple clinical studies have demonstrated that APBI, particularly after breast-conserving surgery, yields satisfactory local control rates comparable to WBI. This is accompanied by reduced side effects, improved convenience, enhanced quality of life, and potential cost savings.

Traditionally, APBI has been administered after surgery, but there is a recent trend to explore preoperative APBI. The rationale for performing preoperative APBI includes several considerations. Firstly, compared to postoperative APBI, the precise location of visually identifiable tumors allows for more accurate and targeted radiation therapy, minimizing the impact on adjacent normal tissues and achieving superior cosmetic results. Secondly, reducing the size of the preoperative lesion may enable more conservative surgery, decreasing the extent of the surgical procedure. Thirdly, it can serve as a preparatory treatment to assess tumor responsiveness. Fourthly, in some cases, it may be administered for definitive purposes, especially in elderly or frail women who may find it challenging to undergo standard treatment due to concurrent health issues.

Several clinical studies have reported the effectiveness and validity of preoperative PBI in a few cases of early breast cancer. These studies have shown low rates of acute and chronic toxicity, with excellent cosmetic outcomes. While accumulating evidence supports preoperative PBI, there is currently a lack of comparative studies with postoperative PBI. Therefore, this study aims to compare and evaluate the overall clinical advantages, including safety and efficacy, of preoperative PBI and postoperative PBI in early breast cancer patients.

DETAILED DESCRIPTION:
This study is a phase II clinical trial consisting of a single experimental group (preoperative PBI group).

- Experimental Group: Preoperative Partial Breast Irradiation (Preoperative PBI)

The objective is to prove that preoperative partial breast irradiation (PBI) is not inferior in terms of radiotherapy-related side effects compared to postoperative PBI in early breast cancer patients.

Treatment outcomes, treatment-related complications, quality of life, degree of breast fibrosis, and breast aesthetics will be prospectively observed. Up to 47 patients will be enrolled over a period of 2 years, with a maximum follow-up observation of 1 years.

Evaluation of acute radiotherapy-related complications will be conducted at least once within 2 weeks from the start of radiotherapy. Additional assessments for acute complications and surgery-related complications will be performed at least once after 6 months of radiotherapy. Evaluation of late radiotherapy-related complications will occur 12 months after radiotherapy.

Patient's quality of life will be measured using self-reported questionnaires at (1) before radiotherapy, (2) 6 months after radiotherapy, and (3) 12 months after radiotherapy.

Breast aesthetics assessment using BCCT. Score software will be conducted at (1) before radiotherapy, (2) 6 months after radiotherapy, and (3) 12 months after radiotherapy. Evaluation of breast fibrosis will utilize the Tissue Compliance Meter device at (1) before radiotherapy, (2) 6 months after radiotherapy, and (3) 12 months after radiotherapy.

Preoperative PBI will be administered within 6 weeks of the patient's first registration, and surgery will be performed within 8 to 12 weeks after radiotherapy. Throughout radiotherapy, immediate, post-treatment, and follow-up observations at 6-month to 1-year intervals for up to 1 years will assess complications, surgical outcomes, cosmetic effects, and disease status.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ductal carcinoma in situ (DCIS) and invasive breast cancer.
* Age ≥ 45
* cT1/cN0, tumor size ≤ 2.5cm
* ECOG 0~2 -ER+, HER2-

Exclusion Criteria:

* cN+
* Tumor located too close to the skin or chest wall (within 5 mm)
* With previous treatment history for breast cancer
* Neoadjuvant chemotherapy
* Multicentric disease
* Diffuse microcalcification
* BRCA mutation
* Paget's disease
* In cases where tumor delineation is not achievable on CT/MRI images

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-10-12 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 2 or higher acute toxicities | Within 6 months after the start of radiotherapy
  The grade of toxicities should be evaluated according to CTCAE version 5.0.

SECONDARY OUTCOMES:
Pathologic complete response (CR) rate | At the time of surgery
Rate of any grade acute toxicities | Within 6 months after the start of radiotherapy
Rate of any gade late toxicities | 6 months after the start of radiotherapy
Rate of grade 2 or higher late toxicities | 6 months after the start of radiotherapy
BCCT.core software score | Baseline (before radiotherapy), at 6 months, 12 months after radiotherapy
Change of Quality of life score | Baseline (before radiotherapy), at 6 months, 12 months after radiotherapy
Tissue compliance meter score | Baseline (before radiotherapy), at 6 months, 12 months after radiotherapy
Disease-free survival | 12 months
overall survival | 12 months
breast cancer specific survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yong Bae Kim, Principal Investigator — Department of Radiation Oncology, Yonsei University College of Medicine
Locations (1):
- Department of Radiation Oncology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No